CLINICAL TRIAL: NCT06895330
Title: Virtual Reality Vs. Helfer Skin Tap: Which One is Helping Children Cope with Fear, Anxiety, and Pain During Vaccination?
Brief Title: Effects of Virtual Reality and Helfer Skin Tap During Vaccination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Hatice ERDEM ÖNDER, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MehmetAkifU-SBF-HEÖ-03
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Fear; Anxiety; Satisfaction
Keywords: pain; fear; anxiety; satistaction; virtual reality; helfer skin tap; vaccine
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Personal Satisfaction; Pain

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned to Virtual reality, Helfer skin tap, and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Group (Experimental): A brief orientation regarding the use of the virtual reality headset will be provided to the children. One minute prior to the vaccination procedure, the selected video-either a roller coaster or Formula 1 experience, based on the child's preference-will be initiated through the virtual reality headset. Throughout the procedure, the children will continue to watch the video using the virtual reality headset.
  Interventions: Other: Virtual Reality Group
- Helfer Skin Tap Group (Experimental): The Helfer Skin Tap technique is applied to reduce pain and muscle tension during intramuscular injection by stimulating large nerve fibers through rhythmic tapping. After determining the injection site and preparing the skin with alcohol, the area is tapped for approximately 5 seconds using the dominant hand. The syringe is then held in the dominant hand while a "V" shape is formed with the non-dominant hand to tap the skin firmly three times. On the count of three, the needle is inserted at a 90° angle. After aspiration, the medication is injected slowly while gentle tapping continues to maintain muscle relaxation. The procedure concludes with simultaneous needle withdrawal and a final V-shaped tap to minimize discomfort.
  Interventions: Other: Helfer Skin Tap Group

INTERVENTIONS:
Other: Virtual Reality Group — A brief orientation regarding the use of the virtual reality headset will be provided to the children. One minute prior to the vaccination procedure, the selected video-either a roller coaster or Formula 1 experience, based on the child's preference-will be initiated through the virtual reality headset. Throughout the procedure, the children will continue to watch the video using the virtual reality headset.
  Arms: Virtual Reality Group
Other: Helfer Skin Tap Group — The Helfer Skin Tap technique is applied to reduce pain and muscle tension during intramuscular injection by stimulating large nerve fibers through rhythmic tapping. After determining the injection site and preparing the skin with alcohol, the area is tapped for approximately 5 seconds using the dominant hand. The syringe is then held in the dominant hand while a "V" shape is formed with the non-dominant hand to tap the skin firmly three times. On the count of three, the needle is inserted at a 90° angle. After aspiration, the medication is injected slowly while gentle tapping continues to maintain muscle relaxation. The procedure concludes with simultaneous needle withdrawal and a final V-shaped tap to minimize discomfort.
  Arms: Helfer Skin Tap Group

SUMMARY:
The aim of this study was to detect and compare the effects of Virtual Reality and Helfer Skin Tap methods on pain, fear, anxiety, and satisfaction during the administration of Tetanus-Diphtheria vaccine to school-aged children. This study was an experimental randomized controlled trial. The sample was included 138 children in a family health centers aged 13 years who underwent Tetanus-Diphtheria vaccine. The participants were randomly assigned to Virtual Reality, Helfer Skin Tap, and control groups. Each group included 46 children, of whom 23 were female and 23 were male. The State-Trait Anxiety Inventory, Children's Fear Scale and Visual Analog Scale were used to collect the data.

DETAILED DESCRIPTION:
This research aims to determine effects of Virtual Reality and Helfer Skin Tap methods on pain, fear, anxiety, and satisfaction during the administration of Tetanus-Diphtheria vaccine to school-aged children.

The following hypotheses were determined for the present study. Hypothesis 1. Virtual Reality is effective in reducing pain, fear and anxiety of children and increasing satisfaction during Tetanus-Diphtheria vaccine injection.

Hypothesis 2. Helfer Skin Tap is effective in reducing pain, fear and anxiety of children and increasing satisfaction during Tetanus-Diphtheria vaccine injection.

Hypothesis 3. Virtual Reality is more effective than Helfer Skin Tap in reducing pain, fear and anxiety of children and increasing satisfaction during Tetanus-Diphtheria vaccine injection.

This prospective, randomized controlled study will be conducted in a family health center in Manisa, Turkey, between May 2025 and December 2025. A parallel-group design will be employed, consisting of three arms: Virtual Reality, Helfer Skin Tap, and a control group. The study protocol will be guided by the Consolidated Standards of Reporting Trials (CONSORT) checklist. All procedures will be performed by the same nurse at the designated family health center to ensure standardization.

Children aged 13 years who will undergo tetanus-diphtheria vaccination will be considered eligible for inclusion. Inclusion criteria will include being 13 years of age and conscious (able to communicate). Exclusion criteria will encompass the presence of any physical or psychological condition, the use of analgesics, sedatives, or anticonvulsants within the preceding 24 hours, diagnosis of any chronic or life-threatening disease, and refusal to participate in the Virtual Reality or Helfer Skin Tap interventions during vaccination.

The sample size for the research was determined using G*power 3.0.8 software, and power analysis was conducted. With a 5% error rate, 80% power, and a medium effect size of 0.25 for the 3 groups with 2 repeated factors, it was calculated that 46 children should be taken for each group (Ellis, 2010). Accordingly, the total sample will consist of 138 children.

Eligible children presenting for tetanus vaccination will be randomly assigned to one of the three groups: Virtual Reality, Helfer Skin Tap, or control (conventional injection technique). To control for potential gender-related effects, children will first be stratified by gender and subsequently randomized into the groups using block randomization.

For randomization and to minimize potential bias, group names (Virtual Reality, Helfer Skin Tap, Control) will be written on identical papers and placed into two separate boxes-pink for females and blue for males. Immediately prior to vaccination, each child will draw a paper from the corresponding box to determine their group allocation. This procedure will ensure gender balance across the groups.

Each group will comprise 46 children, with an equal distribution of 23 females and 23 males.

ELIGIBILITY:
Inclusion Criteria:

* 13 years
* being conscious (with the ability to communicate)

Exclusion Criteria:

* having a physical and psychological condition
* taking any analgesics, sedatives, or anticonvulsants in the past 24 hours
* having chronic or life-threatening disease
* refusing the virtual reality or helfer skin tap technique intervention during vaccine injection.

Ages: 13 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2025-05-03 (Estimated); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The Visual Analog Scale (VAS) will be administered immediately prior to and immediately following the vaccination procedure.
  This scale consists of a 10-cm line (0-10 cm or 0-100 mm). The 0-line on the scale indicates "no pain," and the 10-line indicates "unbearable pain." The child is asked to mark the place that expresses the degree of pain. The distance from the point marked by the child to the 0 line is measured to determine the degree of pain. In children aged 8 and above, the Visual Analog Scale (VAS) is considered the most reliable method.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | State-Trait Anxiety Inventory (STAI) will be administered immediately prior to and immediately following the vaccination procedure.
  The State-Trait Anxiety Inventory (STAI) has been employed in clinical settings to assess levels of both state (STAI-S; i.e., current) and trait (STAI-T; i.e., long-term, general) anxiety. This formwas developed by Spielberger et al. (1971) to measure the anxiety levels of children. The STAI-S was adapted into Turkish by Özusta in 1995, and its validity and reliability study was conducted. The inventory is a 3-point Likert-type scale consisting of 20 items that aim to evaluate feelings associated with state anxiety. The children evaluated how they felt 'at that moment' as "almost never" (1 point), "sometimes" (2 points), and "often" (3 points). The scale ranges from 20 to 60 points, with a high score indicating a high level of anxiety.
Children Fear Scale | Children Fear Scale will be administered immediately prior to and immediately following the vaccination procedure.
  The scale consists of five face shapes scored from 0 to 4. A score of 0 indicates no fear, while a score of 4 indicates serious fear.
Satisfaction level | Satisfaction will be assessed immediately after the vaccination procedure.
  Children will asked to rate their satisfaction level with the vaccination on a scale of 0 points "not satisfied" to 10 points "very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Nihal TASKIRAN, Study Chair — Aydin Adnan Menderes University; Seyma KISLALI TAS, Study Chair — Manisa Soma Family Health Center
Locations (1):
- Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No